CLINICAL TRIAL: NCT03397992
Title: Low Dialysate Temperature to Prevent Intradialytic Hypotension During SLED in AKI
Brief Title: Low Dialysate Temperature During SLED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Fahad Edrees, Principal Investigator, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 201612031
Record Dates: First submitted 2018-01-02; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Acute Kidney Injury; Intra-dialytic Hypotension
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patients, primary providers, ICU nurses and primary nephrology team are blinded. The PI and the dialysis nurses are not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Treatment with high dialysate temperature first followed by low dialysate temperature and alternating thereafter.
  Interventions: Other: Changing dialysate temperature
- Group B (Active Comparator): Treatment with low dialysate temperature first followed by high dialysate temperature and alternating thereafter
  Interventions: Other: Changing dialysate temperature

INTERVENTIONS:
Other: Changing dialysate temperature — Patients had SLED with low dialysate temperature (around 35°C) compared with high dialysate temperature (around 37°C)

SUMMARY:
Objectives: This study is evaluating the hemodynamic effects of lowering the dialysate temperature in acute kidney injury (AKI) patients submitted to sustained low efficiency dialysis (SLED) in a single large center.

Methods: Participants will be randomly assigned to two treatment groups. One group will be started treatment with low temperature (set point 5 on the machine which is around 35°C) for one treatment and then alternate between high and low temperatures for a maximum of 8 treatments. The other group will be started with high temperature (set point 9 on the machine which is around 37°C) for the first treatment then alternate between high and low temperatures for a maximum of 8 treatments. Each participants will need at least two treatments, one with each temperature to be included in the analysis. The investigators will be looking for the number of events during a SLED treatment. Events will be defined as drop in systolic blood pressure ≥ 20 mmHg or drop in mean arterial pressure (MAP) of ≥10 mmHg, requirement of resuscitation with IVF after initiation of SLED, initiation or increase requirement of vasoactive drugs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, AKI stage 3 requiring RRT, maximum two pressers, initial temperature of 36°C or higher.

Exclusion Criteria:

* Initial temperature less than 36°C, ESRD, three or more pressers, requirement of antihypertensive medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-04-22 (Actual); Study Completion 2017-04-22 (Actual)

PRIMARY OUTCOMES:
Number of intradialytic hypotension episodes with different dialysate temperatures | Participants who are enrolled are monitored during SLED treatment which can run from 8 to 14 hours for maximum of 8 treatments or till participant is switched to a different dialysis modality
  Hypothesis is that low dialysate temperature will decrease the number of hypotensive episodes during SLED treatment, hypotensive episodes are defined as drop in SBP ≥ 20 mm Hg or MAP ≥ 10 mm Hg, decrease in ultrafiltration rate, increase or start of vasoactive agents or termination of treatment because of hypotension.

SECONDARY OUTCOMES:
Effect on baseline body temperature | Participants who are enrolled are monitored during SLED treatment which can run from 8 to 14 hours for maximum of 8 treatments or till participant is switched to a different dialysis modality
  Change of body temperature during and at end of SLED treatment from baseline temperature measured before starting SLED
Effect on total ultrafiltration | Participants who are enrolled are monitored during SLED treatment which can run from 8 to 14 hours for maximum of 8 treatments or till participant is switched to a different dialysis modality
  The total amount of fluid ordered to be removed will be compared with the amount actually removed
Effect on Kt/V | Participants who are enrolled are monitored during SLED treatment which can run from 8 to 14 hours for maximum of 8 treatments or till participant is switched to a different dialysis modality
  The dialysis dose will be monitored

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edrees FY, Katari S, Baty JD, Vijayan A. A Pilot Study Evaluating the Effect of Cooler Dialysate Temperature on Hemodynamic Stability During Prolonged Intermittent Renal Replacement Therapy in Acute Kidney Injury. Crit Care Med. 2019 Feb;47(2):e74-e80. doi: 10.1097/CCM.0000000000003508. PMID 30394919